CLINICAL TRIAL: NCT01678014
Title: Phase 1 Study of Deep Brain Stimulation and Capsulotomy for the Treatment of Refractory Anorexia
Brief Title: Deep Brain Stimulation and Capsulotomy for the Treatment of Refractory Anorexia Nervosa
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Wei Liu, Principal Investigator, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DBSAN
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Anorexia
Keywords: Anorexia; DBS; Capsulotomy; Signs and Symptoms
MeSH Terms: conditions — Anorexia; Signs and Symptoms | interventions — Deep Brain Stimulation; Posterior Capsulotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anorexia (Experimental): Anorexia patients
  Interventions: Procedure: Deep Brain Stimulation(DBS); Procedure: Capsulotomy

INTERVENTIONS:
Procedure: Deep Brain Stimulation(DBS) — Deep Brain Stimulation(DBS)is a neurosurgical procedure which include the implantation of deep brain electrodes and the connect to an implantable pulse generator (IPG) that is implanted below the collarbone.
Procedure: Capsulotomy

SUMMARY:
Anorexia nervosa (AN) is a serious eating disorder mostly affecting adolescent girls and young adult women. There are many methods in the treatment of AN, such as family therapy, cognitive behavioral therapy, psychotherapy and so on. However, almost 50% of patients are refractory to all current medical treatment and never fully recover and the standardized mortality ratio over the first 10 years is about 10%. For treatment-refractory anorexia, stereotactic functional neurosurgery may be the better choice. Deep brain stimulation and capsulotomy are the most used methods which has been proved effective in obsessive and compulsive disorders, depression and other psychiatric disorders. Many case reports indicate that deep brain stimulation or capsulotomy may be effective in the treatment of AN. As there are some common pathways between AN and other psychiatric disorder. The investigators have a hypothesis that deep brain stimulation and capsulotomy may be promising methods in the treatment of AN.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a serious eating disorder mostly affecting adolescent girls and young adult women. Although the etiology of AN is still unclear, it is unanimous that social, genetic and psychological factors appear to be involved in the onset and maintenance of this disorder. There are many methods in the treatment of AN, such as family therapy, cognitive behavioral therapy, psychotherapy and so on. However, almost 50% of patients are refractory to all current medical treatment and never fully recover and the standardized mortality ratio over the first 10 years is about 10%. For treatment-refractory anorexia, stereotactic functional neurosurgery may be the better choice. Neurosurgery has been used in the treatment of mental diseases for more than fifty years. Deep brain stimulation and capsulotomy are the most used methods which has been proved effective in obsessive and compulsive disorders, depression and other psychiatric disorders. Many case reports indicate that deep brain stimulation or capsulotomy may be effective in the treatment of AN. As there are some common pathways between AN and other psychiatric disorders. The investigators have a hypothesis that deep brain stimulation and capsulotomy may be promising methods in the treatment of AN.

ELIGIBILITY:
Inclusion Criteria:

1. The age was between 18 to 60 years old.
2. Diagnosis of Anorexia Nervosa by the Diagnostic and Statistical Manual (DSM-IVR)
3. Able to comply with all testing, follow-ups and study appointments and protocols.
4. Treatment Resistance is defined by some or all of:

   * The duration of AN was more than 3 years and no period of good function.
   * The disorder severely affected the quality of life of the patient, preventing participation in normal activities such as work or study.
   * Chronic stable AN lasting at least 10 years.

Exclusion Criteria:

1. Patients with obviously encephalatrophy which was confirmed by MRI.
2. Patients who were alcohol or substance dependence or abuse in the last 6 months.
3. Patients who can not undergo the Magnetic Resonance Imaging (MRI) or Positron Emission Tomography (PET) scanning
4. patients can not complete the 12 months follow-up.
5. Patients with severe heart diseases or other organic problem who could not undergo the neurosurgery.
6. Pregnancy

   -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Anorexia Related Preoccupations and Rituals | April 2012-April 2014
  Change from baseline in Anorexia Related Preoccupations and Rituals scores at 3 months, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bomin Sun, MD, Study Director — Department of sterotactic and functional neurosurgery, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China